CLINICAL TRIAL: NCT05583513
Title: Evaluation of the Progression of Disease and Health-related Quality of Life in Ambulatory Heart Failure Patients: A Local Clinic-based Registry
Brief Title: Heart Failure Evaluation Study
Status: Completed | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, GuangMing Tan, Professor, Chinese University of Hong Kong
Other Study IDs: 2022.204
Record Dates: First submitted 2022-09-26; First posted 2022-10-17 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Heart Failure
Keywords: Heart failure; HF with reduced ejection fraction; HF with preserved ejection fraction; HF exacerbation; quality of life
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Ambulatory Heart Failure
  Interventions: Diagnostic Test: MLHFQ (Minnesota Living with Heart Failure Questionnaire); Diagnostic Test: KCCQ (the Kansas City Cardiomyopathy Questionnaire)

INTERVENTIONS:
Diagnostic Test: MLHFQ (Minnesota Living with Heart Failure Questionnaire) — The MLHFQ, a 21-item HF-specific questionnaire, was adopted to evaluate the quality of life of the study subjects with score ranging 0-105 and lower the scores the better QoL
Diagnostic Test: KCCQ (the Kansas City Cardiomyopathy Questionnaire) — The KCCQ, is a 23-item self-administered questionnaire developed to independently measure the patient's perception of their health status, with score ranging 1-100 and higher scores the better QoL

SUMMARY:
Heart failure (HF) is a highly prevalent conditions that impose a significant burden to the patients, the hospital and the healthcare system. In Hong Kong, HF was one of the commonest causes of hospitalization and death. While HF with reduced ejection fraction (HFrEF) infer high mortality, HF with preserved ejection fraction (HFpEF) can be equally debilitating with similar hospital readmission rate and decline in functional status. Despite recent advancement and approval of novel pharmacologic agents and device therapies to treat HF, HF remains difficult to manage, with increased mortality and frequent hospitalization. HF is characterized by a gradual progression with intervals of exacerbation that often necessitating frequent re-admission. These readmissions are common with up to 1 quarter of patients readmitting within 30 days and half within 6 months8. An ambulatory HF centre can serve both as a transition of care from inpatients to community setting and as a point-of-care for early HF exacerbation (HFE) to prevent recurrent HF hospitalization. This is a registry study aims to investigate the progression disease and its impact on the quality of life (QoL) of the patients who are managed at the ambulatory HF clinic.

DETAILED DESCRIPTION:
Patient population and study location All patients managed at the Prince of Wales Hospital Ambulatory Heart Failure clinic will be recruited into this registry. Patients' consent will be sought from either the patients or their legal guardian should the patients deemed incapable to consent. There are no exclusion criteria.

Collectable Data Patients' demographic information, clinical characteristic including co-morbidities and physical findings, medication records, laboratory parameter including basic blood test and cardiac enzymes which include NT-pro BNP level, imaging parameters including echocardiographic findings and other relevant cardiac imaging findings will be recorded at baseline and at every visit. Patients' functional class as measure by the New York Heart Association (NYHA) classification and their 6 minute walk test will be recorded at selected time point. Patient's Health-related Quality of Life will be measured using both the Minnesota Living with Heart Failure Questionaire (MLHFQ) and the Kansas City Cardiomyopathy Questionnaire (KCCQ) at selected time-point. The MLHFQ, a 21-item HF-specific questionnaire, was adopted to evaluate the quality of life of the study subjects with score ranging 0-105 and lower the scores the better QoL. The KCCQ, is a 23-item self-administered questionnaire developed to independently measure the patient's perception of their health status, with score ranging 1-100 and higher scores the better QoL. All subjects will have the Chinese version of the questionnaire administered by research team at baseline, 3-month and 12-month.

Intervention Since this is a registry, no active intervention will be provided. Treatment of HF will be dictated by the responsible physician.

Duration This registry aim to follow patients for long term.

Analysis All statistical analysis will be performed using STATA version 15 software (College Station, TX, USA). Continuous variables were described by using descriptive statistics including means, medians, and SDs. Frequencies were used for categorical variables. The prevalence of use of each drug was expressed as the percentage of patients using the drug. Wilcoxon Signed Rank Test was performed to test for statistical significance of the differences in NYHA, KCCQ-12 and MLHFQ scores at 3-month and 12-month with respect to the baseline. Kaplan-Meier survival analysis will be performed for time to first hospital admission and death, with time censored at death or on last follow-date. The effect of clinical categories on time to first hospitalization was assessed using adjusted Cox proportional hazards models. Repeat hospitalization outcomes were examined using Cox regression analysis for recurrent events, accounting for the possibility of multiple readmissions occurring over time in the same patient. We treat death and hospitalization as separate competing events. The lifetime of the HF patient is defined to begin on the first registration to the clinic. The MLHFQ-21 and KCCQ-12 domain and summary scores were analysed as continuous variables and grouped scores categories for analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Subject age >18 receiving management at the Ambulatory Heart Failure Clinic

Exclusion Criteria:

1. Subject is unable or unwilling to provide written consent prior to enrollment

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population is base on the primary objective
Sampling Method: Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2023-10-01 (Actual)

PRIMARY OUTCOMES:
Time to first rehospitalization | Change from time to first rehospitalization at 12-months
100 patient-year readmission rate | Change from 100 patient-year readmission rate at 12-months
Change in functional class as measured by NYHA class over times | Change from functional class as measured by NYHA class over times at 12-months
  Class I - No symptoms and no limitation in ordinary physical activity, e.g. shortness of breath when walking, climbing stairs etc.
  Class II - Mild symptoms (mild shortness of breath and/or angina) and slight limitation during ordinary activity.
  Class III - Marked limitation in activity due to symptoms, even during less-than-ordinary activity, e.g. walking short distances (20-100 m).Comfortable only at rest.
  Class IV - Severe limitations. Experiences symptoms even while at rest. Mostly bedbound patients.
  No NYHA class listed or unable to determine.
Change in QoL as measured by MLHFQ and KCCQ over times | Change from QoL as measured by MLHFQ over times at 12-months
  The MLHFQ, a 21-item HF-specific questionnaire, was adopted to evaluate the quality of life of the study subjects with score ranging 0-105 and lower the scores the better QoL.
  The KCCQ, is a 23-item self-administered questionnaire developed to independently measure the patient's perception of their health status, with score ranging 1-100 and higher scores the better QoL.
Change in QoL as measured by KCCQ over times | Change from QoL as measured by KCCQ over times at 12-months
  The KCCQ, is a 23-item self-administered questionnaire developed to independently measure the patient's perception of their health status, with score ranging 1-100 and higher scores the better QoL.
Heart-failure related mortality | Change from Heart-failure related mortality at 12-months

SECONDARY OUTCOMES:
Change in number of Participants With Abnormal Laboratory Values | Change from number of Participants With Abnormal Laboratory Values at 12-months
Change in patients' laboratory parameters | Change from patients' laboratory parameters at 12-months
Change from baseline in log-transformed NT-proBNP level over time | Change from baseline in log-transformed NT-proBNP level over time at 12-months
Change in 6MWT | Change from 6MWT at 12-months
Change of cardiovascular medications | Change of cardiovascular medications at 12-months
  Change of cardiovascular medications, including ACEI/ARB/ARNI, Beta-blockers, Calcium Channel Blockers, Diuretics, Aldosterone antagonist, antiplatelet, anticoagulation, anti-arrythmias, vasodilators, lipid-lowering agents, potassium supplements, SGLT2 inhibitors.
Cardiovascular and All-cause mortality | Change from cardiovascular and All-cause mortality at 12-months
The costs of all services, medications and tests | Change from costs of all services, medications and tests at 12-months
  The costs of all services, medications and tests as estimated with reference to the Hong Kong Government Gazette 2020 and Hong Kong Hospital Authority Drug Formulary 2020

CONTACTS AND LOCATIONS:
Locations (1):
- Prince of Wales Hospital, Hong Kong, Shatin, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Arora S, Lahewala S, Hassan Virk HU, Setareh-Shenas S, Patel P, Kumar V, Tripathi B, Shah H, Patel V, Gidwani U, Deshmukh A, Badheka A, Gopalan R. Etiologies, Trends, and Predictors of 30-Day Readmissions in Patients With Diastolic Heart Failure. Am J Cardiol. 2017 Aug 15;120(4):616-624. doi: 10.1016/j.amjcard.2017.05.028. Epub 2017 Jun 1. PMID 28648393
- [Result] Virani SS, Alonso A, Aparicio HJ, Benjamin EJ, Bittencourt MS, Callaway CW, Carson AP, Chamberlain AM, Cheng S, Delling FN, Elkind MSV, Evenson KR, Ferguson JF, Gupta DK, Khan SS, Kissela BM, Knutson KL, Lee CD, Lewis TT, Liu J, Loop MS, Lutsey PL, Ma J, Mackey J, Martin SS, Matchar DB, Mussolino ME, Navaneethan SD, Perak AM, Roth GA, Samad Z, Satou GM, Schroeder EB, Shah SH, Shay CM, Stokes A, VanWagner LB, Wang NY, Tsao CW; American Heart Association Council on Epidemiology and Prevention Statistics Committee and Stroke Statistics Subcommittee. Heart Disease and Stroke Statistics-2021 Update: A Report From the American Heart Association. Circulation. 2021 Feb 23;143(8):e254-e743. doi: 10.1161/CIR.0000000000000950. Epub 2021 Jan 27. PMID 33501848
- [Result] Savarese G, Lund LH. Global Public Health Burden of Heart Failure. Card Fail Rev. 2017 Apr;3(1):7-11. doi: 10.15420/cfr.2016:25:2. PMID 28785469
- [Result] Reddy YNV, Rikhi A, Obokata M, Shah SJ, Lewis GD, AbouEzzedine OF, Dunlay S, McNulty S, Chakraborty H, Stevenson LW, Redfield MM, Borlaug BA. Quality of life in heart failure with preserved ejection fraction: importance of obesity, functional capacity, and physical inactivity. Eur J Heart Fail. 2020 Jun;22(6):1009-1018. doi: 10.1002/ejhf.1788. Epub 2020 Mar 9. PMID 32150314
- [Result] McDonagh TA, Metra M, Adamo M, Gardner RS, Baumbach A, Bohm M, Burri H, Butler J, Celutkiene J, Chioncel O, Cleland JGF, Coats AJS, Crespo-Leiro MG, Farmakis D, Gilard M, Heymans S, Hoes AW, Jaarsma T, Jankowska EA, Lainscak M, Lam CSP, Lyon AR, McMurray JJV, Mebazaa A, Mindham R, Muneretto C, Francesco Piepoli M, Price S, Rosano GMC, Ruschitzka F, Kathrine Skibelund A; ESC Scientific Document Group. 2021 ESC Guidelines for the diagnosis and treatment of acute and chronic heart failure. Eur Heart J. 2021 Sep 21;42(36):3599-3726. doi: 10.1093/eurheartj/ehab368. No abstract available. PMID 34447992
- [Result] Writing Committee; Maddox TM, Januzzi JL Jr, Allen LA, Breathett K, Butler J, Davis LL, Fonarow GC, Ibrahim NE, Lindenfeld J, Masoudi FA, Motiwala SR, Oliveros E, Patterson JH, Walsh MN, Wasserman A, Yancy CW, Youmans QR. 2021 Update to the 2017 ACC Expert Consensus Decision Pathway for Optimization of Heart Failure Treatment: Answers to 10 Pivotal Issues About Heart Failure With Reduced Ejection Fraction: A Report of the American College of Cardiology Solution Set Oversight Committee. J Am Coll Cardiol. 2021 Feb 16;77(6):772-810. doi: 10.1016/j.jacc.2020.11.022. Epub 2021 Jan 11. No abstract available. PMID 33446410
- [Result] Chun S, Tu JV, Wijeysundera HC, Austin PC, Wang X, Levy D, Lee DS. Lifetime analysis of hospitalizations and survival of patients newly admitted with heart failure. Circ Heart Fail. 2012 Jul 1;5(4):414-21. doi: 10.1161/CIRCHEARTFAILURE.111.964791. Epub 2012 May 2. PMID 22556322
- [Result] Greene SJ, Mentz RJ, Felker GM. Outpatient Worsening Heart Failure as a Target for Therapy: A Review. JAMA Cardiol. 2018 Mar 1;3(3):252-259. doi: 10.1001/jamacardio.2017.5250. PMID 29387880
- [Result] DeVore AD, Allen LA, Eapen ZJ. Thinking Outside the Box: Treating Acute Heart Failure Outside the Hospital to Improve Care and Reduce Admissions. J Card Fail. 2015 Aug;21(8):667-73. doi: 10.1016/j.cardfail.2015.05.009. Epub 2015 May 22. PMID 26009012
- [Result] Zsilinszka R, Mentz RJ, DeVore AD, Eapen ZJ, Pang PS, Hernandez AF. Acute Heart Failure: Alternatives to Hospitalization. JACC Heart Fail. 2017 May;5(5):329-336. doi: 10.1016/j.jchf.2016.12.014. Epub 2017 Mar 8. PMID 28285117
- [Result] Hung YT, Cheung NT, Ip S, Fung H. Epidemiology of heart failure in Hong Kong, 1997. Hong Kong Med J. 2000 Jun;6(2):159-62. PMID 10895138
- [Result] Green CP, Porter CB, Bresnahan DR, Spertus JA. Development and evaluation of the Kansas City Cardiomyopathy Questionnaire: a new health status measure for heart failure. J Am Coll Cardiol. 2000 Apr;35(5):1245-55. doi: 10.1016/s0735-1097(00)00531-3. PMID 10758967
- See also: HA Statistical Report — https://www3.ha.org.hk/data/HAStatistics/StatisticalReport/